CLINICAL TRIAL: NCT06366841
Title: Stigma and Psychological profilE in REctal-anal caNcer pAtients
Acronym: SERENA
Status: Recruiting | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: 6439
Record Dates: First submitted 2024-04-05; First posted 2024-04-16 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Rectal Cancer; Anal Cancer
MeSH Terms: conditions — Rectal Neoplasms; Anus Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Psychological tests administration — Psychological tests administration to evaluate stigma, personality characteristics and quality of life of rectal and anal cancer patients.

SUMMARY:
In 2022, Italy is estimated to have 48,100 cases of colon-rectum cancer. Locally advanced mid-lower rectal cancers require preoperative chemo-radiotherapy with fluoropyrimidine. The diagnosis and treatment of rectal cancer have a significant impact on patients' well-being, causing physical and psychological distress. Symptoms such as abdominal pain, fatigue, diarrhea, are commonly reported. While distress levels have been examined before, the relationship between other aspects of the patient experience, such as psychosocial factors, stigma, temperament and personality, alexithymia, have not been extensively explored. Colorectal cancer is associated with specific socially stigmatized challenges. Stigmatization is defined as societal identification of an individual as abnormal and worthy of separation, leading to discrimination and loss of social status. Rectal cancer patients may perceive high levels of stigma and blame due to factors such as defecation-related symptoms, colonoscopy or rectal examinations, physical limitations, loss of work ability and the use of colostomy or ileostomy. Anal cancer, although traditionally surrounded by social stigma, is gaining awareness worldwide due to increasing diagnoses. In other forms of cancer, stigma has been linked to personality traits. Given the characteristics related to the illness and the profile of rectal and anal cancer patients, it is important to assess the psychological traits and psychological resources, also in order to establish tailored psychological pathways during the disease trajectory that comprehend chemoradiations and possible subsequent surgery. Currently, there is no documented data on the relationship between stigma, and psychological profiles in rectal and anal cancer patients. Aim of this protocol is to evaluate the stigma, and psychopathological profile in rectal and anal cancer patients and to evaluate changes in those variables over time.

ELIGIBILITY:
Inclusion Criteria:

Locally advanced rectal and anal cancer patients undergoing a long course of radiotherapy

* Patients in chemo-radiation treatment
* Ability to understand and complete the questionnaires
* Age ≥18 years
* Informed consent signed

Exclusion Criteria:

* Age > 75 years
* Rectal and anal cancer patients undergoing short-course radiotherapy
* Rectal and anal cancer patients undergoing palliative radiotherapy
* Patients with inability to express informed consent
* Patients denying informed consent
* Patients with psychopathological disturbances preexisting to the cancer diagnosis
* Patients affected by severe language deficits

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Rectal and anal cancer patients undergoing a long course of radiotherapy
Sampling Method: Probability Sample
Enrollment: 148 (Estimated)
Dates: Start 2024-05-06 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Evaluation of rectal and anal cancer stigma | 24 months
  PSS (modified) Perceived Stigma Scale. A self-administered questionnaire to measure perceived stigma through 7 items on a five-point Likert scale (ranging from 0 = never to 4 = always), with a higher score reflecting a greater level of perceived stigma (min score 0 max score 28).

SECONDARY OUTCOMES:
Evaluation of psychological characteristics in rectal and anal cancer | 24 months
  Personality Inventory for DSM-5 (Diagnostic Statistical Manual of Mental Disorders 5th edition) brief form for adults The Personality Inventory for DSM-5 brief form measures non-adaptive personality traits: Negative Affectivity, Detachment, Antagonism, Disinhibition and Psychoticism (25 items).
Temperament Evaluation of Memphis, Pisa, Paris and San Diego-autoquestionnaire brief version | 24 months
  Temperament Evaluation of Memphis, Pisa, Paris and San Diego-autoquestionnaire brief version. is a new self-report measure of the affective temperament with depressive (D), cyclothymic (C), hyperthymic (H), irritable (I), and anxious (A) subscales.
Toronto Alexithymia Scale | 24 months
  Alexithymia Toronto Scale is a 20-item Likert scale. Within the TAS, there are distinct subscales that focus on specific dimensions of alexithymia: Difficulty Describing Feelings, Difficulty Identifying Feelings, and Externally Oriented Thinking.
EORTC QLQ - CR29 and EORTC QLQ-ANL27 | 24 months
  EORTC QLQ - CR29 and EORTC QLQ-ANL27 Quality of life in rectal and anal cancer submodules specifically assess colon-rectal and anal cancer. Raw scores for each scale are linear transformed into a 0-100 outcome. A higher functioning score indicated better functioning or global health/QoL, whereas higher symptom scores indicate a higher level of symptom severity.

CONTACTS AND LOCATIONS:
Overall Officials: Loredana Dinapoli, Principal Investigator — Fondazione Policlinico Universitario A. Gemelli, IRCCS
Locations (2):
- Italy (2):
  - Fondazione Policlinico Universitario A. Gemelli IRCCS - Psychology service, Roma
  - Fondazione Policlinico Universitario A. Gemelli IRCCS, Roma